CLINICAL TRIAL: NCT07360652
Title: Acute Effects of an Elastic Band Rewarm-Up Protocol on Vertical Jump Performance in Highly Trained Female Volleyball Players: a Crossover Study
Brief Title: Effects of an Elastic Band Rewarm-Up in Highly Trained Female Volleyball Players
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University Institute of Maia (Other)
Responsible Party: Principal Investigator, Henrique Sousa, Principal Investigator, University of Maia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: EBT_HS_04
Record Dates: First submitted 2025-12-09; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Physical Performance Parameters

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Elastic bands rewarm-up (Experimental): Rewarm-up with elastic bands
  Interventions: Other: EB RWU
- CG (No Intervention): No rewarm-up

INTERVENTIONS:
Other: EB RWU — Rewarm-up with elastic bands
  Arms: Elastic bands rewarm-up

SUMMARY:
This study aims to examine the acute effects of an elastic band rewarm-up on vertical jump performance in highly trained female volleyball players. A randomized crossover design will be used, with participants completing three sessions. Session 1 will serve as a familiarization with the testing and the rewarm-up protocol. In Sessions 2 and 3, participants will be divided into two groups. Group 1 will perform a standard warm-up followed by 5 minutes of rest, then an elastic band rewarm-up, while Group 2 will perform the warm-up followed by 5 minutes of rest only. In the subsequent session, the protocols will be crossed over so that each participant completes both conditions. Vertical jump performance will be assessed using the Chronojump system, evaluating both countermovement jumps (CMJ) and Abalakov jumps. To mimic real-game conditions, athletes will rotate between the vertical jump evaluations and simulated match play, allowing investigation of the acute effects of an elastic band rewarm-up on explosive lower-limb performance during volleyball-specific activity.

ELIGIBILITY:
Inclusion Criteria:

* belong to the U-21 or Senior level of a women's volleyball club.
* be apart of a national volleyball championship

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Biologically Female
Enrollment: 30 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Vertical Jump | The evaluations will be conducted at baseline (before the warm-up), immediately after the warm-up intervention, after the 5 minute rest, and after 4 minutes, 8 minutes and 12 minutes of the simulated match.
  Jump height and power will be evaluated using Chronojump system, evaluating both countermovement jumps (CMJ) and Abalakov jumps. The players will perform the CMJ, where they will begin from an upright position, with their hands on their hips; a rapid downward movement to a knee angle of ∼90°, immediately transitioning to propel themselves upwards into the air. The abalakov jump is similar to the CMJ; the only difference is that the hands can move freely while jumping.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maia, Maia, Porto District, Portugal

IPD SHARING:
Plan to Share IPD: Undecided